CLINICAL TRIAL: NCT02655562
Title: Fractional Concentration of Exhaled NO(FeNO) to Direct The Treatment of Sub-acute Cough：A Prospective, Open Label, Randomized and Placebo-Controlled Trial
Brief Title: Fractional Concentration of Exhaled NO(FeNO) to Direct The Treatment of Sub-acute Cough
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: There are difficulties in recruiting patients
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Mingming Jiang, Principal Investigator, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing Chao Yang Hospital
Record Dates: First submitted 2015-12-30; First posted 2016-01-14 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Coughing
MeSH Terms: conditions — Cough | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- biomarker treatment arm (Experimental): Patients in biomarker treatment arm and FENO≥25ppb were given Montelukast Sodium Tablets (p.o., 10mg, qd) . Patients in biomarker reatment arm and FENO<25ppb were given placebo (p.o., 10mg, qd).All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Interventions: Drug: Montelukast
- standard treatment arm (Placebo Comparator): Patients in standard treatment arm and FENO≥25ppb were given placebo (p.o., 10mg, qd). Patients in standard treatment arm and FENO<25ppb were given Montelukast Sodium Tablets (p.o., 10mg, q.d.).All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Patients in biomarker treatment arm and FENO≥25ppb were given Montelukast Sodium Tablets (p.o., 10mg, qd) . Patients in biomarker reatment arm and FENO<25ppb were given placebo (p.o., 10mg, qd).
  Patients in standard treatment arm and FENO≥25ppb were given placebo (p.o., 10mg, qd). Patients in standard treatment arm and FENO<25ppb were given Montelukast Sodium Tablets (p.o., 10mg, q.d.).All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Other Names: Placebo

SUMMARY:
Cough is a common symptom that leads patients worldwide to seek medical attention. Subacute cough refers to a cough of 3-8-week duration, and is typically refractory to standard anti-tussive therapy, and a tendency to spontaneous healing was common. Few clinical trials have evaluated therapeutic options for subacute cough. Airway inflammation is an important feature of most of subacute cough, Cysteinyl leukotrienes and FeNO correlates with airway inflammation. Subacute cough often represents a prolonged post-viral response. Cysteinyl leukotrienes increase in virus infection. Airway inflammation induce epithelial cells produce iNOS(inducible nitric oxide synthase,iNOS), and FeNO increase in theory. Montelukast is a cysteinyl leukotriene type 1 receptor antagonist that is reported to improve cough16 and reduces FENO and prevents increases in FENO during reduction of inhaled corticosteroid dose, But A meta-analysis of the effectiveness of LTRA( leukotriene receptor antagonist,LTRA)in treating children with prolonged non-specific cough concluded that, with the lack of evidence, the routine use of LTRA in treating children with non-specific cough cannot be recommended. A randomised, placebo-controlled trial showed montelukast is not an effective treatment for postinfectious cough. Non-specialists or general practitioners of Japan prescribe LTRA very often, which increase. The aim is to research whether FeNO can be used as a biomarker to direct montelukast treatment and optimize treatment regimen of sub-acute cough.

DETAILED DESCRIPTION:
This project is a prospective, open label, randomized and controlled trial. All subacute cough patients that met the inclusion/exclusion criteria were recruited after signing the consent form. Patients were randomized into biomarker treatment armand standard treatment arm.

Patients in biomarker treatment arm and FENO≥25ppb were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) . Patients in biomarker reatment arm and FENO<25ppb were given placebo (p.o., 10mg, qd). Patients in standard treatment arm and FENO≥25ppb were given placebo (p.o., 10mg, qd). Patients in standard treatment arm and FENO<25ppb were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) .All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.

Examine results of all patients from all arms were recorded before and after the 10 day treatment. The examine recorded are FENO levels, cough symptom assessment, cough visual assessment, Leicester cough questionnaire, total white blood cell count, neutrophil blood percentage, eosinophil blood percentage. Patient cough free days after treatment and Montelukast Sodium Tablets . Follow up was carried out at the 8th week after first record of symptom and 2 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cough is the main or only clinical symptom and was persistent for 3-8 weeks Chest X-ray reveals no noticeable pathological changes
* more than 18 year old, regardless of gender and ethical background
* Not taking angiotensin-converting enzyme inhibitor
* Patients must join the programme voluntarily and are able to attend examination and follow-up sessions

Exclusion Criteria:

* Patients diagnosed with allergic rhinitis, chronic nasosinusitis or bacterial respiratory tract infections
* Patients diagnosed with severe reportorial disease of other severe systemic disease
* Patients who are allergic to any drugs to be tested
* Patients who are non-cooperative during examination sessions or other steps of the trial
* Patients who are not able to or refuse to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2024-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Leicester cough questionnaire | 10 days
  Change in Leicester Cough Questionnaire(LCQ) total and domain scores at 10 days post randomisation

SECONDARY OUTCOMES:
cough visual assessment | 10 days
  Change in Leicester Cough Questionnaire(LCQ) physical,psychological and social domain scores at 10 days post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Kewu Huang, M.D., Study Chair — Respiratory Medicine Department
Locations (1):
- Mingming Jiang, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wedde-Beer K, Hu C, Rodriguez MM, Piedimonte G. Leukotrienes mediate neurogenic inflammation in lungs of young rats infected with respiratory syncytial virus. Am J Physiol Lung Cell Mol Physiol. 2002 May;282(5):L1143-50. doi: 10.1152/ajplung.00323.2001. PMID 11943681
- [Background] van Schaik SM, Tristram DA, Nagpal IS, Hintz KM, Welliver RC 2nd, Welliver RC. Increased production of IFN-gamma and cysteinyl leukotrienes in virus-induced wheezing. J Allergy Clin Immunol. 1999 Apr;103(4):630-6. doi: 10.1016/s0091-6749(99)70235-6. PMID 10200012
- [Background] Spector SL, Tan RA. Effectiveness of montelukast in the treatment of cough variant asthma. Ann Allergy Asthma Immunol. 2004 Sep;93(3):232-6. doi: 10.1016/S1081-1206(10)61493-7. PMID 15478381
- [Background] Kato A, Schleimer RP. Beyond inflammation: airway epithelial cells are at the interface of innate and adaptive immunity. Curr Opin Immunol. 2007 Dec;19(6):711-20. doi: 10.1016/j.coi.2007.08.004. Epub 2007 Oct 24. PMID 17928212
- [Background] Mincheva RK, Kralimarkova TZ, Rasheva M, Dimitrov Z, Nedeva D, Staevska M, Papochieva V, Perenovska P, Bacheva K, Dimitrov VD, Popov TA. A real - life observational pilot study to evaluate the effects of two-week treatment with montelukast in patients with chronic cough. Cough. 2014 Mar 20;10(1):2. doi: 10.1186/1745-9974-10-2. PMID 24649919
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Background] Sandrini A, Ferreira IM, Gutierrez C, Jardim JR, Zamel N, Chapman KR. Effect of montelukast on exhaled nitric oxide and nonvolatile markers of inflammation in mild asthma. Chest. 2003 Oct;124(4):1334-40. doi: 10.1378/chest.124.4.1334. PMID 14555563
- [Background] Wang K, Birring SS, Taylor K, Fry NK, Hay AD, Moore M, Jin J, Perera R, Farmer A, Little P, Harrison TG, Mant D, Harnden A. Montelukast for postinfectious cough in adults: a double-blind randomised placebo-controlled trial. Lancet Respir Med. 2014 Jan;2(1):35-43. doi: 10.1016/S2213-2600(13)70245-5. Epub 2013 Dec 2. PMID 24461900
- [Result] Kwon NH, Oh MJ, Min TH, Lee BJ, Choi DC. Causes and clinical features of subacute cough. Chest. 2006 May;129(5):1142-7. doi: 10.1378/chest.129.5.1142. PMID 16685003
- [Result] Lim KG, Mottram C. The use of fraction of exhaled nitric oxide in pulmonary practice. Chest. 2008 May;133(5):1232-42. doi: 10.1378/chest.07-1712. PMID 18460522
- [Result] Tarnoky AL. Albumin. Ann Clin Biochem. 1981 Mar;18 (Pt 2):61-3. doi: 10.1177/000456328101800201. No abstract available. PMID 7259071
- [Result] Sato S, Saito J, Sato Y, Ishii T, Xintao W, Tanino Y, Ishida T, Munakata M. Clinical usefulness of fractional exhaled nitric oxide for diagnosing prolonged cough. Respir Med. 2008 Oct;102(10):1452-9. doi: 10.1016/j.rmed.2008.04.018. Epub 2008 Jul 9. PMID 18614345
- [Result] Tamaoki J, Kondo M, Sakai N, Nakata J, Takemura H, Nagai A, Takizawa T, Konno K. Leukotriene antagonist prevents exacerbation of asthma during reduction of high-dose inhaled corticosteroid. The Tokyo Joshi-Idai Asthma Research Group. Am J Respir Crit Care Med. 1997 Apr;155(4):1235-40. doi: 10.1164/ajrccm.155.4.9105060.
- [Result] Morice AH, Fontana GA, Sovijarvi AR, Pistolesi M, Chung KF, Widdicombe J, O'Connell F, Geppetti P, Gronke L, De Jongste J, Belvisi M, Dicpinigaitis P, Fischer A, McGarvey L, Fokkens WJ, Kastelik J; ERS Task Force. The diagnosis and management of chronic cough. Eur Respir J. 2004 Sep;24(3):481-92. doi: 10.1183/09031936.04.00027804. No abstract available. PMID 15358710
- [Result] Gentile DA, Fireman P, Skoner DP. Elevations of local leukotriene C4 levels during viral upper respiratory tract infections. Ann Allergy Asthma Immunol. 2003 Sep;91(3):270-4. doi: 10.1016/S1081-1206(10)63529-6. PMID 14533659
- [Result] Grant CC. Postinfectious cough and pertussis in primary care. Lancet Respir Med. 2014 Jan;2(1):2-3. doi: 10.1016/S2213-2600(13)70260-1. Epub 2013 Dec 2. No abstract available. PMID 24461880
- [Result] Dahlen SE. Treatment of asthma with antileukotrienes: first line or last resort therapy? Eur J Pharmacol. 2006 Mar 8;533(1-3):40-56. doi: 10.1016/j.ejphar.2005.12.070. Epub 2006 Feb 28. PMID 16510137
- [Result] Dicpinigaitis PV. Cough: an unmet clinical need. Br J Pharmacol. 2011 May;163(1):116-24. doi: 10.1111/j.1476-5381.2010.01198.x. PMID 21198555